CLINICAL TRIAL: NCT05357157
Title: Effect of Electroacupuncture Treatment on Pain, Mechanical Hyperalgesia, Quality of Life and Expression of Mu+ B Cells in Patients With Fibromyalgia: A Prospective Observational Study
Brief Title: Electroacupuncture Pain Treatment, Mechanical Hyperalgesia, Quality of Life & Expression of Mu+ B Cells in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: University of Crete (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Emmanouela Koutoulaki, Principal investigator, University of Crete
Other Study IDs: Acupuncture - Fibromyalgia
Record Dates: First submitted 2022-01-11; First posted 2022-05-02 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Fibromyalgia; Electroacupuncture; Acupuncture; Hyperalgesia
Keywords: Fibromyalgia; Chronic Pain; Electroacupuncture; Acupuncture; Palmitoylethanolamide; MOR-Positive B Cell; Hyperalgesia; Quality of life; Pressure Algometry; Anti-inflammatory Nutrition; Depression
MeSH Terms: conditions — Fibromyalgia; Hyperalgesia; Chronic Pain; Depression | interventions — Electroacupuncture; Nutritional Status; Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken from patients at the following time periods:
  1. Before the 1st session of electroacupuncture
  2. after the 12th session of electroacupuncture
  3. 6 months after the last session of electroacupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electroacupuncture: All subjects will be administered electroacupuncture sessions Acupoints that will be used: Baihui, Yin tang, BL-10, GB21, SI13, BL-60, ST-36, LV-3, LV8, Spl 6, LI-4, LI11, Kid 3, Ren 6, Heart 7
  Interventions: Other: Electroacupuncture
- Electroacupuncture, Nutrition and Dietary supplement: All subjects will be administered electroacupuncture sessions Acupoints that will be used: Baihui, Yin tang, BL-10, GB21, SI13, BL-60, ST-36, LV-3, LV8, Spl 6, LI-4, LI11, Kid 3, Ren 6, Heart 7. Patients will be presented with the option to be prescribed a dietary supplement containing vitamin B complex, Mg, Zn, superoxide dismutase, Alpha Lipoic Acid and PalmitoylethanolamideAdditionally they will be given a specific anti-intiflamatory dietary regimen to follow.
  Interventions: Other: Electroacupuncture; Dietary Supplement: Nutrition; Dietary Supplement: Dietary supplement

INTERVENTIONS:
Other: Electroacupuncture — Subjects will be administered electroacupuncture as described in the electroacupuncture group description
Dietary Supplement: Nutrition — Subjects will be administered the intervention described in the electroacupuncture nutrition and dietary supplement group description
  Groups: Electroacupuncture, Nutrition and Dietary supplement
Dietary Supplement: Dietary supplement — Subjects will be administered the intervention described in the electroacupuncture nutrition and dietary supplement group description
  Groups: Electroacupuncture, Nutrition and Dietary supplement

SUMMARY:
Fibromyalgia (FM) is a complex, multifactorial syndrome characterized by widespread chronic pain with hyperal- gesia and allodynia and a constellation of somatic and psychological manifestations, including fatigue, sleep dis- orders, depression, anxiety, gastrointestinal and cognitive disorders. FM is now recognized as one of the most common chronic pain conditions and its management remains a challenge for patients and healthcare profes- sionals. The fact that FM is associated with chronic pain without any obvious peripheral tissue damage has given rise to the concept of nociplastic pain with evidence of dysfunction in mono-aminergic neurotransmission, lead- ing to elevated levels of excitatory neurotransmitters and decreased levels of serotonin and norepinephrine in the spinal cord at the level of descending anti-nociceptive pathways. Additionally, dopamine dysregulation and altered activity of endogenous cerebral opioids have been observed in FM.

Recent European guidelines on FM treatment emphasize that there should be a comprehensive assessment of patient's pain, function and psychosocial context. It is recognized that there are profound and fundamental problems associated with the pain assessment tools in common use, as most of these represent an attempt to reduce a multidimensional experience to a coarse unidimensional measure. Use of multiple tools for sub- jective and objective assessment of pain may reflect more accurately patient's pain experience. Furthermore, tracing a biologic pain marker in FM patients would facilitate both the initial assessment of pain and the re- sponse to treatment. Management of pain in FM patients should focus first on non-pharmacological modalities. Acupuncture therapy is an effective and safe treatment and exerts its analgesic effect through activation of pe- ripheral and central pain control systems with the release of β-endorphins, enkephalins, dynorphins, serotonin, norepinephrine, γ-aminobutyric acid or ATP. The aim of our study is to assess initially reported pain and evaluate the effectiveness of electroacupuncture (with or without diet modifications) on the "whole experience of pain" in FM patients in a multimodel assessment frame.

DETAILED DESCRIPTION:
The International Association for the Study of Pain (IASP) defined chronic pain as pain that persists or recurs for more than three months. In the case of conditions such as FM, it can be conceived as a disease in its own, right de- scribed as "chronic primary pain", and the existence of such persisting pain, despite adequate treatment and in the absence of any sign of inflammation, has led researchers to look for evidence of central sensitization.

Misuse and misreporting of chronic pain assessment run deep, both in research and the clinical setting. Chronic pain diagnosis lacks specific tools to objectively define pathology, unlike other diseases (e.g., oncology or infectiol- ogy), where biomarkers play a well-known role. The objectivity of pain severity is still described only in terms of pain threshold and patients have to rate their pain considering a numeric rating scale (NRS) of 0 to 10, where zero is a no pain condition and a 10 means the pain is as bad as it could be, even if it involves many other factors, such as anthropological, spiritual, genetic, social, and psychological personal experience.

Currently, there is no internationally accepted classification of pain severity for FM and the physician is tasked with careful evaluation in order to determine the most effective treatment. It is common practice to consider a '30% reduction' in pain reported in verbal numerical rating scores (VNRS) as adequate pain response to treatment. This is problematic for several reasons. While there have been arguments for and against the linearity of a properly ad- ministered VAS there is no adequate evidence that a VNRS can be treated as linear, nor that any given score repre- sents the same thing from one individual to another or indeed from one day to another even for any given individ- ual. The use of a mean to summarize VNRS data is therefore likely to be inappropriate, as would be the application of parametric statistics to those data, although this is perhaps more controversial if the samples are very large. For the same reason, it is not appropriate to quantify a percent reduction in pain from such a study. Given the multidi- mensional and very individual nature of the pain experience, the concept of quantifying any alteration in pain as a percentage does not seem appropriate.

The American College of Rheumatology (ACR) criteria for FM diagnosis have changed over time, maintaining ad- vantages and limitations and clinicians rely only on clinical examination and questionnaire administration to make a diagnosis. Neither specific diagnostic laboratory tests nor biomarkers are available to confirm FM diagnosis, espe- cially in its specificity of chronic widespread pain (CWP). Little is known about the role of opioid receptors on circu- lating cells during the development of a chronic pain disease. In recent years, attention has been focused on the close association between peripheral nerve and opioid-containing immune cells. Both immune cells and neurons share common ligands and receptors, and this ligand-receptor communication influences and activates cellular path- ways in both systems. The complex communication between endogenous antinociceptive systems, pathology and peripheral opioid receptors has encouraged a hypothesis that lymphocyte opioid Mu receptor (MOR) expression could serve as a biomarker for FM diagnosis and pain assessment. In a recent study, the percentage of Mu-positive B cells was investigated as a biological marker for an objective diagnosis of chronic pain suffering patients, also con- tributing to the legitimacy of FM as a truly painful disease. . In the study by Raffaeli et al, it was certi- fied that FM pain perception is an objective widespread chronic pain status where pain is the primary symptom and FM pathogenesis derives from a characteristic morphological modulation of the endogenous antinociceptive path- way. It was suggested that a lower expression of Mu+ B cells in FM patients seemed to be linked to a reduced thresh- old level of pain response and that a low availability of opioid receptors in FM patients could show altered endoge- nous opioid analgesic activity.

A multimodel assessment model of pain incorporates pain experience, pain expression, and pain measures. The aim of our study is to evaluate the effectiveness of electroacupuncture on the "whole" pain experience and quality of life in FM patients with the use of multiple tools; in addition to a patient's self-reported value on a numerical scale for the assessment of pain will be used:

1. measurement of percentage of Mu + B-lymphocytes in a blood sample (biological marker)
2. assessment of pressure pain thresholds with the use of an algometer
3. PSD scale for monitoring the severity of fibromyalgia symptoms
4. quality of life questionnaire in patients with fibromyalgia
5. Detection of depression with a questionnaire (Patient health questionnaire, PHQ-9) It is the first time that mu-receptor (MOR) expression in B lymphocytes will be used as biomarker of pain re- sponse to treatment in patients with fibromyalgia undergoing electro-acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient's consent
* Age >18 years old
* Patients with diagnosed fibromyalgia from rheumatologists
* Widespread pain more than 6 months
* In case of drug therapy, it should be taken at least one month before the beginning of the session and remain stable till the end of the study

Exclusion Criteria:

* Deep depression
* Biological agent use ( TNF inhibitors)
* Heamatological diseases
* Systemic Infections
* pregnancy
* electroacupuncture contraindications (epilepsy, pacemaker/ implantable cardioverter defibrillator (ICD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be referred from Rheumatology clinic with an established primary fibromyalgia diagnosis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
MOR - positive Bcells - baseline | Baseline
  Patients' blood samples will be collected prior to the intervention to serve as a baseline. Flow cytometry immunophenotyping will be performed on the samples to determine the percentage of MOR positive B cells. Data will be reported as a percentage of the total B cell number.
MOR - positive Bcells - 6th session of electroacupuncture | End of 6th session of electroacupuncture- 3 weeks after baseline
  Patients' blood samples will be collected at the end of the 6th session of electroacupuncture. All patients will undergo electroacupuncture sessions twice a week, and the first 6 electroacupuncture sessions will take place within 3 weeks. Flow cytometry immunophenotyping will be performed on the samples to determine the percentage of MOR positive B cells. Data will be reported as a percentage of the total B cell number.
MOR - positive Bcells - 12th session of electroacupuncture | End of 12th session of electroacupuncture - 6 weeks after baseline
  Patients' blood samples will be collected at the end of the 12th session of electroacupuncture. All patients will undergo electroacupuncture sessions twice a week, and all 12 electroacupuncture sessions will take place within 6 weeks. Flow cytometry immunophenotyping will be performed on the samples to determine the percentage of MOR positive B cells. Data will be reported as a percentage of the total B cell number.
MOR - positive Bcells - 6 months after the end of the 12th session | 6 months after the end of 12th session of electroacupuncture
  Patients' blood samples will be collected 6 months after the end of the 12th session of electroacupuncture. All patients will undergo electroacupuncture sessions twice a week, and all 12 electroacupuncture sessions will take place within 6 weeks. Patients will undergo no more electroacupuncture sessions after the 12th session. Flow cytometry immunophenotyping will be performed on the samples to determine the percentage of MOR positive B cells. Data will be reported as a percentage of the total B cell number.

SECONDARY OUTCOMES:
Pain estimation with Pressure algometer - baseline (trapezius) | baseline
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the trapezius muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - baseline (supraspinatus) | baseline
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the supraspinatus muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - baseline (tibia) | baseline
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the tibia bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 6th session of electroacupuncture (trapezius) | end of 3rd week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the trapezius muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 6th session of electroacupuncture (supraspinatus) | end of 3rd week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the supraspinatus muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 6th session of electroacupuncture (tibia) | end of 3rd week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the tibia bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - end of 12th session of electroacupuncture (trapezius) | end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the trapezius muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - end of 12th session of electroacupuncture (supraspinatus) | end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the supraspinatus muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - end of 12th session of electroacupuncture (tibia) | end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the tibia bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 3 months after the end of the 12th electroacupuncture session(trapezius) | 3 months after the end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the trapezius muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 3 months after the end of the 12th electroacupuncture session(supraspinatus) | 3 months after the end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the supraspinatus muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 3 months after the end of the 12th electroacupuncture session(tibia) | 3 months after the end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the tibia bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 6 months after the end of the 12th electroacupuncture session(trapezius) | 6 months after the end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the trapezius muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 6 months after the end of the 12th electroacupuncture session(supraspinatus) | 6 months after the end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the supraspinatus muscle bilaterally and the mean value will be reported.
Pain estimation with Pressure algometer - 6 months after the end of the 12th electroacupuncture session(tibia) | 6 months after the end of 6th week of electroacupuncture
  Patients will undergo Pressure pain threshold estimation with a pressure algometer. Measurements will be taken at the tibia bilaterally and the mean value will be reported.
Pain evaluation - baseline | baseline
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Pain evaluation - after the end of 6th session | end of 3rd week of electroacupuncture
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Pain evaluation - after the end of 12th session | after the end of 6th week of electroacupuncture
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Pain evaluation - 3 months after the end of 12th session | 3 months after the end of 6th week of electroacupuncture
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Pain evaluation - 6 months after the end of 12th session | 6 months after the end of 6th week of electroacupuncture
  Evaluation of patients' pain using scales: Numerical Rating Scale (NRS). The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
PHQ-9 (Patient Health Questionnaire-9) - baseline | baseline
  Patients will fill in a standardized questionnaire (PHQ-9). Results will be reported on a 0 - 27 scale
PHQ-9 (Patient Health Questionnaire-9) - after the end of 6th session | after the end of 3rd week of electroacupuncture
  Patients will fill in a standardized questionnaire (PHQ-9). Results will be reported on a 0 - 27 scale
PHQ-9 (Patient Health Questionnaire-9) - after the end of 12th session | after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (PHQ-9). Results will be reported on a 0 - 27 scale
PHQ-9 (Patient Health Questionnaire-9) - 3 months after the end of 12th session | 3 months after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (PHQ-9). Results will be reported on a 0 - 27 scale
PHQ-9 (Patient Health Questionnaire-9) - 6 months after the end of 12th session | 6 months after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (PHQ-9). Results will be reported on a 0 - 27 scale
Fibromyalgia Impact Questionnaire Score-Revised (FIQ-R) - baseline | baseline
  Patients will fill in a standardized questionnaire (FIQ-R). Results will be reported on a 0 - 100 scale.
Fibromyalgia Impact Questionnaire Score-Revised (FIQ-R) - after the end of 6th session | after the end of 3rd week of electroacupuncture
  Patients will fill in a standardized questionnaire (FIQ-R). Results will be reported on a 0 - 100 scale.
Fibromyalgia Impact Questionnaire Score-Revised (FIQ-R) - after the end of 12th session | after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (FIQ-R). Results will be reported on a 0 - 100 scale.
Fibromyalgia Impact Questionnaire Score-Revised (FIQ-R) - 3 months after the end of 12th session | 3 months after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (FIQ-R). Results will be reported on a 0 - 100 scale.
Fibromyalgia Impact Questionnaire Score-Revised (FIQ-R) - 6 months after the end of 12th session | 6 months after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (FIQ-R). Results will be reported on a 0 - 100 scale.
Polysymptomatic Distress Scale (PDS) - baseline | baseline
  Patients will fill in a standardized questionnaire (PDS). Results will be reported on a 0 - 31 scale.
Polysymptomatic Distress Scale (PDS) - after the end of 6th session | after the end of 3rd week of electroacupuncture
  Patients will fill in a standardized questionnaire (PDS). Results will be reported on a 0 - 31 scale.
Polysymptomatic Distress Scale (PDS) - after the end of 12th session | after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (PDS). Results will be reported on a 0 - 31 scale.
Polysymptomatic Distress Scale (PDS) - 3 months after the end of 12th session | 3 months after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (PDS). Results will be reported on a 0 - 31 scale.
Polysymptomatic Distress Scale (PDS) - 6 months after the end of 12th session | 6 months after the end of 6th week of electroacupuncture
  Patients will fill in a standardized questionnaire (PDS). Results will be reported on a 0 - 31 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heraklion, Heraklion, Greece